CLINICAL TRIAL: NCT06493955
Title: Evaluation of the Effectiveness of Extending the "Passerelle" System for Prescribing Adapted Physical Activity to Patients With Type 2 Diabetes in Nouvelle-AQUItaine (France)
Acronym: PAPA-NAQUI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2023/47
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Adapted Physical Activity; general practice
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: comparative, multicenter, interventional, superiority study, randomized in two unblinded parallel groups. Randomization will be 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Patients with type 2 diabetes included in the adapted physical activity arm for 12 months
  Interventions: Other: Adapted physical activity for 12 months
- control arm (Active Comparator): Type 2 diabetes patients with standard prescription for adapted physical activity (6 months)
  Interventions: Other: Adapted physical activity for 6 months

INTERVENTIONS:
Other: Adapted physical activity for 12 months — 6 additional months of adapted physical activity after the 6 first months
  Arms: experimental arm
Other: Adapted physical activity for 6 months — standard 6-month prescription for adapted physical activity
  Arms: control arm

SUMMARY:
Type 2 diabetes is on the increase worldwide. Two major risk factors have been identified: overweight and physical inactivity. National and international recommendations encourage general practitioner to guide patients in changing their lifestyle. As regards physical activity in France, general practitioner have been able to prescribe adapted physical activity (APA) for their patients since 2016. In type 2 diabetes, it is known that physical activity interventions are cost-effective. However, these interventions are often too expensive and far removed from real life. It is also known that the benefits of intervention increase up to 18 months, then diminish to zero at 36 months. In Nouvelle-Aquitaine, France, the "PEPS Sport-santé network", offers physical activity coaching for patients who are not sufficiently active: the "Passerelle" program. Patients can benefit from a weekly physical activity session for 6 months.

The investigators would therefore like to assess whether extending the existing "Passerelle program" by 6 months, with one session every 15 days, is effective in maintaining the volume of physical activity 12 months after the end of the intervention.

DETAILED DESCRIPTION:
Over the last few decades, we have witnessed an increasing rise in the prevalence of chronic diseases, including type 2 diabetes (T2DM). Internationally, diabetes affected 108 million people in the 1980s, compared with 451 million in 2017, reaching epidemic proportions according to the World Health Organization (WHO). France has not been spared by T2DM, with an estimated prevalence of 11.8% in 2017 and an incidence of 10.7 cases per 1,000 person-years. The chronic hyperglycemia of type 2 diabetes is associated with altered macronutrient metabolism, with a lack of insulin secretion or reduced insulin sensitivity. Insulin resistance impairs the ability of muscle cells to absorb and store glucose. Two major modifiable risk factors have been identified: overweight and physical inactivity. T2DM increases the risk of myocardial infarction and stroke by a factor of 2 to 3. The ENTRED 3 study carried out in 2019 among diabetic patients in mainland France showed that 18.6% of type 2 diabetic patients had had a coronary complication and 7.8% a stroke. In addition to these two macro-vascular complications, diabetes is responsible for micro-vascular complications such as retinopathy and diabetic nephropathy. The cost to society of physical inactivity is considerable. Worldwide, healthcare expenditure linked to T2DM and physical inactivity has been estimated at 37.6 billion dollars.

The management of type 2 diabetic patients aims to reduce morbidity and mortality through glycemic control. The latest French recommendations for the management of diabetic patients date from 2014, and encourage doctors to monitor their patients every three months to ensure compliance, look for risk factors and comorbidities (hypertension, smoking and alcohol consumption), measure blood pressure, weight and calculate BMI. HbA1c tests should be carried out between two and four times a year. The first recommended hypoglycemic treatment is based on physical activity and diet.

More recent recommendations from the American Diabetes Association (ADA) in 2022 encourage physicians to manage patients using a multifactorial approach. First-line management involves lifestyle changes, promoting healthier behaviors around diet, physical activity promotion, substance use such as smoking, weight loss and sleep quality.

Sport-health networks such as the PEPS network in the Nouvelle-Aquitaine region (Prescription d'Exercice Physique pour la Santé - Prescription of Physical Exercise for Health) make it easier for patients to be referred to a suitable structure for supervised exercise.

Investigators would like to know whether extending this program with spaced sessions can encourage patients to change their behavior over the long term. Spacing out the sessions should enable a smoother transition to independent or associative practice.

The research question is as follows: What is the effectiveness of a one-year Passerelle program in maintaining the volume of physical activity in T2DM patients in the Nouvelle-Aquitaine region?

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes with initial diagnosis of fasting blood glucose > 1.26 g/l on 2 occasions
* Patient aged 18 or over
* Patient with a Marshall score ≤ 3
* Patient residing in the Nouvelle-Aquitaine region
* Patient eligible for the "Passerelle" program
* Patient willing to participate
* Patient agreeing to take part in the study and having signed an informed consent form
* Person affiliated or benefiting from a social security scheme.

Exclusion Criteria:

* Patient with any other unstabilized pathology:
* Cardiovascular: unstable angina, stress angina, malignant hypertension, recent myocardial infarction, unstabilized heart disease
* Pulmonary: uncontrolled asthma, COPD exacerbation
* Endocrine: diabetes with HbA1c > 9%, plantar perforator disease
* Pregnant patient
* Diabetic patient with contraindication to APA prescription
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
ONAPS-PAQ questionnaire, | 12 months after the end of the intervention
  Measurement of weekly physical activity volume using the " national observatory on physical activity and sedentariness - physical activity questionnaire" (ONAPS-PAQ), score given in minutes per week : under 150 min/week : Higher early mortality risk, associated with a sharp increase in the risk of chronic diseases above 150min/week : reduced risk of early mortality risk of developing chronic diseases

SECONDARY OUTCOMES:
Physical activity | Month 0 (inclusion) and Month 6, Month 12, Month 18, Month 24 after inclusion
  changes in physical activity volume at baseline and then every 6 months until the end of the study
Sedentariness | At inclusion and 6 months after inclusion and 12 months after the end of the intervention.
  ONAPS PAQ sedentariness score :
  score in minutes of activity : under 150 min/week : Higher early mortality risk, associated with a sharp increase in the risk of chronic diseases above 150min/week : reduced risk of early mortality risk of developing chronic diseases
Weight change | At inclusion and 6 months after inclusion and 12 months after the end of the intervention.
  Difference in weight change between the two groups
Walk test | At inclusion and 6 months after inclusion and 12 months after the end of the intervention.
  6-minute walk test
Therapeutic escalation | 12 months after the end of the intervention.
  Difference in therapeutic escalation level between the two groups
HbA1c | At inclusion and 6 months after inclusion and 12 months after the end of the intervention.
  Difference in HbA1c between the two groups
Quality of life (SF-36) | At inclusion and 6 months after inclusion and 12 months after the end of the intervention.
  Difference in quality of life score between the two groups, measured by the SF-36 quality of life scale.
  The SF-36 scale ranges from 0 to 100. A low score reflects a perception of poor health, loss of function and the presence of pain. A high score reflects a perception of good health, absence of functional deficit and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet Médical Bergerac, Bergerac, France